CLINICAL TRIAL: NCT05062876
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of AD-214 to AD-2141 in Healthy Volunteers
Brief Title: A Study to Compare PK, PD and Safety of the AD-214 and AD-2141
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-214PK/PD-03
Record Dates: First submitted 2021-09-22; First posted 2021-09-30 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-10

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-T (Active Comparator): Period 1 : Test Drug(AD-214) Period 2 : Reference Drug(AD-2141)
  Interventions: Drug: AD-214; Drug: AD-2141
- T-R (Active Comparator): Period 1 : Reference Drug(AD-2141) Period 2 : Test Drug(AD-214)
  Interventions: Drug: AD-214; Drug: AD-2141

INTERVENTIONS:
Drug: AD-214 — 1 tablet administered before the breakfast during 7 days
  Other Names: Test drug
Drug: AD-2141 — 1 tablet administered before the breakfast during 7 days
  Other Names: Reference Drug

SUMMARY:
A study to compare safety, pharmacokinetics and pharmacodynamics of AD-214 to AD-2141 in healthy volunteers.

DETAILED DESCRIPTION:
This study is to compare the safety, pharmacokinetic characteristics and pharmacodynamics characteristics of AD-214 compared with administration of AD-2141 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~50 years in healthy volunteers
* BMI is more than 18.0 kg/m^2 , no more than 27.0 kg/m^2
* Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss(Area under the plasma drug concentration-time curve) | From Day 1 up to Day 29
  Evaluateion PK Rabeprazole after multiple dose
Gastric acidity(After 7days of repeated administration, The change of integrated gastric acidity) | Day1 24hours pH monitoring, Day7 24hours pH monitoring, Day22 24hours monitoring, Day28 24hours pH monitoring
  Evaluation PD Rabeprazole after multiple dose

SECONDARY OUTCOMES:
AUCtau(Area under the plasma drug concentration-time curve) | Day1
  Evaluation PK Rabeprazole after single dose
Cmax(Maximum concentration of drug in plasma) | Day1
  Evaluation PK Rabeprazole after single dose
Tmax(Time to maximum plasma concentration) | Day1
  Evaluation PK Rabeprazole after single dose
t1/2(Terminal elimination half-life) | Day1
  Evaluation PK Rabeprazole after single dose
CL/F(Apparent clearance) | Day1
  Evaluation PK Rabeprazole after single dose
Vd/F(Apparent volume of distribution) | Day1
  Evaluation PK Rabeprazole after single dose
Cmax,ss(Maximum concentration of drug in plasma at steady state) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
Cmin,ss(Minimum concentration of drug in plasma at steady state) Cmin,SS(Minimum concentration of drug in plasma) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
Cav,ss(Average concentration of drug in plasma at steady state) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
Tmax,ss(Time to maximum plasma concentration at steady state) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
t1/2,ss(Terminal elimination half-life at steady state) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
CLss/F(Apparent Clearance at steady state) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
Vss/F(Apparent Volume of distribution at steady state) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
PTF(Peak trough fluctuation over one dosing interal at steady state) | From Day 1 up to Day 29
  Evaluation PK Rabeprazole after multiple dose
After the first administration of esomeprazole, The change of integrated gastric acidity compared to baseline for 24 hours | Day1 24hours monitoring
  Evaluation PD Rabeprazole
After the first dose and 7 days of repeated dosing, Percentage of time to maintain gastric pH 4.0 or higher for 24 hours | Day1 24hours pH monitoring, Day7 24hours pH monitoring, Day22 24hours monitoring, Day28 24hours pH monitoring
  Evaluation PD Rabeprazole
After the first administration and 7 days of repeated administration, The median pH measured for 24 hours | Day1 24hours pH monitoring, Day7 24hours pH monitoring, Day22 24hours monitoring, Day28 24hours pH monitoring
  Evaluation PD Rabeprazole

CONTACTS AND LOCATIONS:
Overall Officials: Seunghwan Lee, M.D.,Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No